CLINICAL TRIAL: NCT04485104
Title: An Open-label, Single-arm Study to Assess the Safety, Pharmacokinetics, and Efficacy of Adjunctive Cannabidiol Oral Solution (GWP42003-P) in Participants With Tuberous Sclerosis Complex (Age 1 Month to < 2 Years of Age), Dravet Syndrome (1 Year to < 2 Years of Age), or Lennox-Gastaut Syndrome (1 Year to < 2 Years of Age) Who Experience Inadequately-controlled Seizures
Brief Title: Assessment of Adjunctive Cannabidiol Oral Solution (GWP42003-P) in Children With Tuberous Sclerosis Complex (TSC), Dravet Syndrome (DS), or Lennox-Gastaut Syndrome (LGS) Who Experience Inadequately-controlled Seizures
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated by the Sponsor due to low patient enrollment.
Sponsor: Jazz Pharmaceuticals (Industry)
Collaborators: Jazz Pharmaceuticals Research UK Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GWEP17005; 2020-002132-67 (EudraCT Number)
Record Dates: First submitted 2020-07-21; First posted 2020-07-24 (Actual); Results first posted 2025-10-31 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Seizure in Participants With Tuberous Sclerosis Complex; Seizure in Participants With Dravet Syndrome; Seizure in Participants With Lennox-Gastaut Syndrome
Keywords: Epilepsy; Seizures; Infantile Spasms; Pediatric; Children; Infants; Cannabidiol oral solution; GWP42003-P; Tuberous Sclerosis Complex; TSC; Tuberous Sclerosis; Cannabidiol; Epidiolex; CBD; Seizure; Child; TSC1; TSC2; Tuberous Sclerosis 1; Tuberous Sclerosis 2; Lennox-Gastaut Syndrome; Dravet Syndrome
MeSH Terms: conditions — Epilepsy; Seizures; Spasms, Infantile; Tuberous Sclerosis; Tuberous Sclerosis 1; Tuberous Sclerosis 2; Lennox Gastaut Syndrome; Epilepsies, Myoclonic | interventions — Cannabidiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- GWP42003-P (Experimental): The 52-week treatment period includes a fixed 2-week titration schedule followed by flexible dose optimization.
  Day 1: 5 mg/kg/day (2.5 mg/kg twice daily (b.i.d.))
  Day 8: 10 mg/kg/day (5 mg/kg b.i.d.)
  Day 15 to Week 52: Flexible dosing based on the participant's observed efficacy, safety, and tolerability per the investigator's clinical judgement. Up to a maximum of 20 mg/kg/day (10 mg/kg b.i.d.) for LGS and DS or 25 mg/kg/day (12.5 mg/kg b.i.d.) for TSC, in maximum weekly increments of 5 mg/kg/day (≤ 2.5 mg/kg b.i.d.).
  Interventions: Drug: GWP42003-P

INTERVENTIONS:
Drug: GWP42003-P — Oral Solution
  Other Names: Cannabidiol; Epidiolex; Epidyolex

SUMMARY:
This study will be conducted to evaluate the safety, pharmacokinetics (PK), and efficacy of adjunctive GWP42003-P in participants < 2 years of age with tuberous sclerosis complex (TSC), Lennox-Gastaut syndrome (LGS), or Dravet syndrome (DS).

DETAILED DESCRIPTION:
The study duration will be up to approximately 62 weeks, including a 4-week screening/baseline period, a 52-week dose optimization treatment period (which includes a fixed 2-week titration period followed by flexible dose optimization), a 10-day taper period, and a safety follow-up period (4 weeks after the end-of-taper visit).

ELIGIBILITY:
Key Inclusion Criteria:

* Participants with TSC (1 month to < 2 years of age), or DS (1 year to < 2 years of age), or LGS (1 year to < 2 years of age) within the specified age range at the time of initial informed consent.
* Parent(s)/legal representative is/are willing and able to give informed consent for participation in the study.
* Parent(s)/legal representative is/are willing and able (in the investigator's opinion) to comply with all study requirements (including accurate electronic participant-reported outcome [ePRO] diary completion).
* Participants with TSC must have a diagnosis per the 2012 International Tuberous Sclerosis Complex Consensus Conference. Participants with LGS or DS must have a diagnosis that is consistent with International League Against Epilepsy (ILAE) guidelines and confirmed by the Epilepsy Study Consortium (ESCI).
* Participants who have uncontrolled seizures, and who are currently receiving 1 or more antiseizure medication (ASMs).
* A suitable VEEG, as available in the medical record, within 1 year of Visit 1. When a historical VEEG is not available, and if clinically indicated and appropriate (due to uncertainties or new seizures), a VEEG will be completed and read to confirm diagnosis prior to Visit 3. All VEEGs are to be read at baseline by the investigator and by an independent reviewer.
* Has seizures which are not adequately controlled through their current ASMs, defined as ≥ 1 seizure reported on the seizure diary during the screening/baseline period

Key Exclusion Criteria:

* Has tumor growth which, in the opinion of the investigator, could affect participant safety.
* Has clinically significant abnormal laboratory values, in the investigator's opinion, at screening/baseline.
* Has clinically significant abnormalities in the electrocardiogram (ECG) measured at screening/baseline.
* Has any concurrent cardiovascular conditions, that will, in the investigator's opinion, interfere with the ability to assess their ECGs.
* Has any known or suspected hypersensitivity to cannabinoids or any of the excipients of the study intervention such as sesame seed oil.
* Has significantly impaired hepatic function prior to Visit 3, defined as:

  * Serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 3 × upper limit of normal (ULN) and (total bilirubin [TBL] > 2 × ULN or international normalized ratio [INR] > 1.5).
  * Serum ALT or AST > 5 × ULN.
  * Serum ALT or AST > 3 × ULN with the presence of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, and/or eosinophilia (> 5%).
  * Elevated ALT or AST should be discussed with the medical monitor prior to Visit 3; the medical monitor may allow for a confirmatory re-draw prior to Visit 3.
* Has received another study intervention within 4 weeks prior to Visit 1 or plans to take another study intervention during the study.
* Has any other clinically significant disease or disorder which, in the opinion of the investigator, may either put the participant, other participants, or site staff at risk because of participation in the study, may influence the result of the study, or may affect the participant's ability to take part in the study.
* Any clinically significant abnormalities identified following a physical examination of the participant that, in the opinion of the investigator, would jeopardize the safety of the participant if they took part in the study.
* Has previously been enrolled into this study.
* Has plans to travel outside their country of residence during the study, unless the participant has confirmation that the study intervention is permitted in the destination country.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 1 Month to 23 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2021-05-19 (Actual); Primary Completion 2025-01-28 (Actual); Study Completion 2025-01-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (6):
  - Clinical Trial Site, Little Rock, Arkansas
  - Clinical Trial Site, Los Angeles, California
  - Clinical Trial Site, Chicago, Illinois
  - Clinical Trial Site, Boston, Massachusetts
  - Clinical Trial Site, Cincinnati, Ohio
  - Clinical Trial Site, Houston, Texas
- Italy (3):
  - Clinical Trial Site, Florence
  - Clinical Trial Site, Genova
  - Clinical Trial Site, Rome
- Spain (2):
  - Clinical Trial Site, Barcelona
  - Clinical Trial Site, Madrid

IPD SHARING:
Plan to Share IPD: Yes
In accordance with ICMJE requirements, Jazz Pharmaceuticals may provide qualified external researchers access to individual participant data (IPD) and clinical trial data that underlie the results of this trial upon request. Qualified researchers can submit a request on https://www.jazzpharma.com/science/clinical-trial-data-sharing/ as outlined. Jazz Pharmaceuticals reserves the right not to consider a request. For inquiries about Jazz's data sharing policy contact clinicaldatasharing@jazzpharma.com.
URL: https://www.jazzpharma.com/science/clinical-trial-data-sharing

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 3 participants who met all inclusion criteria and no exclusion criteria were enrolled in the study at 3 sites in the United States.
Pre-assignment Details: The study duration will be up to approximately 62 weeks, including a 4-week screening/baseline period, a 52-week dose optimisation treatment period (which includes a fixed 2-week titration period followed by flexible dose optimisation), a 10-day taper period, and a safety follow-up period (4 weeks after the end-of-taper visit).
Groups:
- Tuberous Sclerosis Complex: Participants with Tuberous Sclerosis Complex who received GWP42003-P orally twice daily (b.i.d.) on a titration schedule, with a starting dose of 5 mg/kg/day (2.5 mg/kg b.i.d.) on Day 1, then 10 mg/kg/day (5 mg/kg b.i.d.) on Day 8, followed by a flexible dose optimization from Day 15 to Week 52 based on the clinical judgment of the investigator.
- Dravet Syndrome: Participants with Dravet Syndrome who received GWP42003-P orally twice daily (b.i.d.) on a titration schedule, with a starting dose of 5 mg/kg/day (2.5 mg/kg b.i.d.) on Day 1, then 10 mg/kg/day (5 mg/kg b.i.d.) on Day 8, followed by a flexible dose optimization from Day 15 to Week 52 based on the clinical judgment of the investigator.
Period: Overall Study
Arm/Group | Tuberous Sclerosis Complex | Dravet Syndrome
Started | 2 | 1
Completed | 0 | 0
Not Completed | 2 | 1
Not completed — Physician Decision | 2 | 0
Not completed — Decision by sponsor | 0 | 1

BASELINE CHARACTERISTICS:
Population: Demographic characteristics were assessed in the Safety Analysis Set.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tuberous Sclerosis Complex | Dravet Syndrome | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 1 | 3
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Time Frame: From start of treatment to the post-treatment safety follow-up visit, up to 62 weeks
Population: Treatment-emergent adverse events (TEAEs) were assessed in the Safety Analysis Set.
Measure: Number; unit: participants
Arm/Group | Tuberous Sclerosis Complex | Dravet Syndrome
Number analyzed (Participants) | 2 | 1
participants | 2 | 1

2. Primary Outcome: Mean Change From Baseline in Blood Pressure
Time Frame: From baseline up to the end of taper follow-up visit (Visit 20), up to 62 weeks
Population: Blood pressure was assessed in the Safety Analysis Set.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Tuberous Sclerosis Complex | Dravet Syndrome
Number analyzed (Participants) | 2 | 1
mmHg
  Systolic blood pressure | -3.0 (9.90) | 11.0 (NA) — Standard deviation cannot be calculated for 1 person.
  Diastolic blood pressure | 13.5 (19.09) | -2.0 (NA) — Standard deviation cannot be calculated for 1 person.

3. Primary Outcome: Mean Change From Baseline in Pulse Rate
Time Frame: From baseline up to the end of taper follow-up visit (Visit 20), up to 62 weeks
Population: Pulse rate was assessed in the Safety Analysis Set.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Tuberous Sclerosis Complex | Dravet Syndrome
Number analyzed (Participants) | 2 | 1
beats per minute | -11.0 (1.41) | 11.0 (NA) — Standard deviation cannot be calculated for 1 person.

4. Primary Outcome: Mean Change From Baseline in Respiratory Rate
Time Frame: From baseline up to the end of taper follow-up visit (Visit 20), up to 62 weeks
Population: Respiratory rate was assessed in the Safety Analysis Set.
Measure: Mean (Standard Deviation); unit: breaths/minute
Arm/Group | Tuberous Sclerosis Complex | Dravet Syndrome
Number analyzed (Participants) | 2 | 1
breaths/minute | -10.0 (16.97) | 0 (NA) — Standard deviation cannot be calculated for 1 person.

5. Primary Outcome: Mean Change From Baseline in Body Temperature
Time Frame: From baseline up to the end of taper follow-up visit (Visit 20), up to 62 weeks
Population: Body temperature was assessed in the Safety Analysis Set.
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | Tuberous Sclerosis Complex | Dravet Syndrome
Number analyzed (Participants) | 2 | 1
degrees Celsius | -0.05 (0.354) | -0.10 (NA) — Standard deviation cannot be calculated for 1 person.

6. Primary Outcome: Mean Change From Baseline in Height
Time Frame: From baseline up to the end of taper follow-up visit (Visit 20), up to 62 weeks
Population: Height was assessed in the Safety Analysis Set.
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Tuberous Sclerosis Complex | Dravet Syndrome
Number analyzed (Participants) | 2 | 1
centimeters | 1.95 (1.344) | 4.20 (NA) — Standard deviation cannot be calculated for 1 person.

7. Primary Outcome: Mean Change From Baseline in Body Weight
Time Frame: From baseline up to the end of taper follow-up visit (Visit 20), up to 62 weeks
Population: Body weight was assessed in the Safety Analysis Set.
Measure: Mean (Standard Deviation); unit: kilogram
Arm/Group | Tuberous Sclerosis Complex | Dravet Syndrome
Number analyzed (Participants) | 2 | 1
kilogram | 0.15 (0.354) | 0.60 (NA) — Standard deviation cannot be calculated for 1 person.

8. Primary Outcome: Mean Change From Baseline in Heart Rate
Time Frame: From baseline up to the end of taper follow-up visit (Visit 20), up to 62 weeks
Population: Heart rate was assessed in participants with available data in the Safety Analysis Set.
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | Tuberous Sclerosis Complex | Dravet Syndrome
Number analyzed (Participants) | 1 | 1
beats/minute | -10.0 (NA) — Standard deviation cannot be calculated for 1 person. | 8.0 (NA) — Standard deviation cannot be calculated for 1 person.

9. Primary Outcome: Mean Change From Baseline in RR Interval
Time Frame: From baseline up to the end of taper follow-up visit (Visit 20), up to 62 weeks
Population: RR interval was assessed in participants with available data in the Safety Analysis Set.
Measure: Mean (Standard Deviation); unit: millisecond
Arm/Group | Tuberous Sclerosis Complex | Dravet Syndrome
Number analyzed (Participants) | 1 | 1
millisecond | 48.0 (NA) — Standard deviation cannot be calculated for 1 person. | -45.0 (NA) — Standard deviation cannot be calculated for 1 person.

10. Primary Outcome: Mean Change From Baseline in PR Interval
Time Frame: From baseline up to the end of taper follow-up visit (Visit 20), up to 62 weeks
Population: PR interval was assessed in the Safety Analysis Set.
Measure: Mean (Standard Deviation); unit: millisecond
Arm/Group | Tuberous Sclerosis Complex | Dravet Syndrome
Number analyzed (Participants) | 2 | 1
millisecond | 11.0 (12.73) | -2.0 (NA) — Standard deviation cannot be calculated for 1 person.

11. Primary Outcome: Mean Change From Baseline in QRS Duration
Time Frame: From baseline up to the end of taper follow-up visit (Visit 20), up to 62 weeks
Population: QRS duration was assessed in the Safety Analysis Set.
Measure: Mean (Standard Deviation); unit: millisecond
Arm/Group | Tuberous Sclerosis Complex | Dravet Syndrome
Number analyzed (Participants) | 2 | 1
millisecond | 3.0 (1.41) | 6.0 (NA) — Standard deviation cannot be calculated for 1 person.

12. Primary Outcome: Mean Change From Baseline in QT Interval
Time Frame: From baseline up to the end of taper follow-up visit (Visit 20), up to 62 weeks
Population: QT interval was assessed in the Safety Analysis Set.
Measure: Mean (Standard Deviation); unit: millisecond
Arm/Group | Tuberous Sclerosis Complex | Dravet Syndrome
Number analyzed (Participants) | 2 | 1
millisecond | 0 (8.49) | 0 (NA) — Standard deviation cannot be calculated for 1 person.

13. Primary Outcome: Mean Change From Baseline in QTcB and QTcF
Time Frame: From baseline up to the end of taper follow-up visit (Visit 20), up to 62 weeks
Population: QTcB and QTcF were assessed in participants with available data in the Safety Analysis Set.
Measure: Mean (Standard Deviation); unit: millisecond
Arm/Group | Tuberous Sclerosis Complex | Dravet Syndrome
Number analyzed (Participants) | 1 | 1
millisecond
  QTcB | -10.0 (NA) — Standard deviation cannot be calculated for 1 person. | 16.0 (NA) — Standard deviation cannot be calculated for 1 person.
  QTcF | -4.0 (NA) — Standard deviation cannot be calculated for 1 person. | 9.0 (NA) — Standard deviation cannot be calculated for 1 person.

14. Primary Outcome: Number of Participants With a Clinically Significant Change in Laboratory Parameters
Time Frame: From baseline up to the end of taper follow-up visit (Visit 20), up to 62 weeks
Population: Clinically significant change in laboratory parameters were assessed in participants with available data in the Safety Analysis Set.
Measure: Number; unit: participants
Arm/Group | Tuberous Sclerosis Complex | Dravet Syndrome
Number analyzed (Participants) | 2 | 1
participants
  Alanine aminotransferase | 0 | 1
  Aspartate aminotransferase | 0 | 1
  Gamma Glutamyltransferase | 0 | 1

15. Primary Outcome: Number of Participants With Emergence of New Types of Seizures
Time Frame: From baseline up to the end of taper follow-up visit (Visit 20), up to 62 weeks
Population: New types of seizures were assessed in the Safety Analysis Set.
Measure: Number; unit: participants
Arm/Group | Tuberous Sclerosis Complex | Dravet Syndrome
Number analyzed (Participants) | 2 | 1
participants | 1 | 0

16. Primary Outcome: Plasma Concentrations of GWP42003-P and Its Major Metabolites
Time Frame: Predose, 3 hours and 6 hours post dose at End of Treatment (Week 52)
Population: Pharmacokinetics were assessed and reported for participants when samples were collected. For both participants with Tuberous Sclerosis Complex, it was not possible to collect PK samples at 6hr post dose.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Tuberous Sclerosis Complex | Dravet Syndrome
Number analyzed (Participants) | 2 | 1
ng/mL
  CBD (pre-dose) | 55.3 (46.3) | 99.8 (NA) — Standard deviation cannot be calculated for 1 person.
  CBD (3-hour post-dose): number analyzed (Participants) | 1 | 1
  CBD (3-hour post-dose) | 456 (NA) — Standard deviation cannot be calculated for 1 person. | 427 (NA) — Standard deviation cannot be calculated for 1 person.
  CBD (6-hour post-dose): number analyzed (Participants) | 0 | 1
  CBD (6-hour post-dose) |  | 149 (NA) — Standard deviation cannot be calculated for 1 person.
  7-OH-CBD (pre-dose) | 37.8 (29.7) | 123 (NA) — Standard deviation cannot be calculated for 1 person.
  7-OH-CBD (3-hour post-dose): number analyzed (Participants) | 1 | 1
  7-OH-CBD (3-hour post-dose) | 161 (NA) — Standard deviation cannot be calculated for 1 person. | 580 (NA) — Standard deviation cannot be calculated for 1 person.
  7-OH-CBD (6-hour post-dose): number analyzed (Participants) | 0 | 1
  7-OH-CBD (6-hour post-dose) |  | 292 (NA) — Standard deviation cannot be calculated for 1 person.
  7-COOH-CBD (pre-dose) | 2790 (884) | 7460 (NA) — Standard deviation cannot be calculated for 1 person.
  7-COOH-CBD (3-hour post-dose): number analyzed (Participants) | 1 | 1
  7-COOH-CBD (3-hour post-dose) | 4870 (NA) — Standard deviation cannot be calculated for 1 person. | 10700 (NA) — Standard deviation cannot be calculated for 1 person.
  7-COOH-CBD (6-hour post-dose): number analyzed (Participants) | 0 | 1
  7-COOH-CBD (6-hour post-dose) |  | 9680 (NA) — Standard deviation cannot be calculated for 1 person.

17. Primary Outcome: Number of Participants Based on Percentage Change From Baseline in Indication-Specific Total Countable Seizures as Recorded by Caregivers
Time Frame: Day 1 up to Taper Period, up to Week 52
Population: Indication-specific total countable seizures where assessed in the Safety Analysis Set.
Measure: Number; unit: participants
Arm/Group | Tuberous Sclerosis Complex | Dravet Syndrome
Number analyzed (Participants) | 2 | 1
participants
  Day 1-29: > 25% (increase) | 2 | 0
  Day 1-29: >= 0% to <=25% (increase) | 0 | 0
  Day 1-29: > -25% to 0% (reduction) | 0 | 0
  Day 1-29: <= -25% to > -50% change (reduction) | 0 | 1
  Day 1-29: <= -50% to > -75% change (reduction) | 0 | 0
  Day 1-29: <= -75% (reduction) | 0 | 0
  Day 30-57: > 25% (increase) | 0 | 0
  Day 30-57: >= 0% to <=25% (increase) | 1 | 0
  Day 30-57: > -25% to 0% (reduction) | 0 | 0
  Day 30-57: <= -25% to > -50% change (reduction) | 0 | 0
  Day 30-57: <= -50% to > -75% change (reduction) | 0 | 1
  Day 30-57: <= -75% (reduction) | 0 | 0
  Day 58-85: > 25% (increase) | 0 | 0
  Day 58-85: >= 0% to <=25% (increase) | 1 | 0
  Day 58-85: > -25% to 0% (reduction) | 0 | 0
  Day 58-85: <= -25% to > -50% change (reduction) | 0 | 0
  Day 58-85: <= -50% to > -75% change (reduction) | 0 | 0
  Day 58-85: <= -75% (reduction) | 0 | 1
  Day 86-113: > 25% (increase) | 0 | 0
  Day 86-113: >= 0% to <=25% (increase) | 0 | 0
  Day 86-113: > -25% to 0% (reduction) | 0 | 0
  Day 86-113: <= -25% to > -50% change (reduction) | 0 | 0
  Day 86-113: <= -50% to > -75% change (reduction) | 0 | 1
  Day 86-113: <= -75% (reduction) | 1 | 0
  Day 114-141: > 25% (increase) | 0 | 0
  Day 114-141: >= 0% to <=25% (increase) | 0 | 0
  Day 114-141: > -25% to 0% (reduction) | 0 | 0
  Day 114-141: <= -25% to > -50% change (reduction) | 0 | 0
  Day 114-141: <= -50% to > -75% change (reduction) | 0 | 1
  Day 114-141: <= -75% (reduction) | 1 | 0
  Day 142-169: > 25% (increase) | 0 | 0
  Day 142-169: >= 0% to <=25% (increase) | 0 | 0
  Day 142-169: > -25% to 0% (reduction) | 0 | 0
  Day 142-169: <= -25% to > -50% change (reduction) | 0 | 0
  Day 142-169: <= -50% to > -75% change (reduction) | 0 | 0
  Day 142-169: <= -75% (reduction) | 1 | 0
  Day 170-197: > 25% (increase) | 0 | 0
  Day 170-197: >= 0% to <=25% (increase) | 0 | 0
  Day 170-197: > -25% to 0% (reduction) | 0 | 0
  Day 170-197: <= -25% to > -50% change (reduction) | 0 | 0
  Day 170-197: <= -50% to > -75% change (reduction) | 0 | 0
  Day 170-197: <= -75% (reduction) | 1 | 0
  Taper Period: > 25% (increase) | 1 | 0
  Taper Period: >= 0% to <=25% (increase) | 0 | 0
  Taper Period: > -25% to 0% (reduction) | 0 | 0
  Taper Period: <= -25% to > -50% change (reduction) | 0 | 0
  Taper Period: <= -50% to > -75% change (reduction) | 0 | 0
  Taper Period: <= -75% (reduction) | 0 | 0

18. Primary Outcome: Clinician Global Impression of Severity (CGI/S) Score
Description: The CGIC/S is a comprehensive neurodevelopmental assessment that covers the following domains: sensory, motor, cognition, emotional/behavioral health, communication, social, and adaptive functioning. This assessment is a 2-question survey per domain to be completed by the clinician. Individual domain scores are reported.
  The severity of impairment in each domain is rated by the clinician in a scale of 1 through 7 where 1 = Normal, not at all ill; 2 = Borderline ill; 3 = Mildly ill; 4 = Moderately ill; 5 = Markedly ill; 6 = Severely ill; 7 = Among the most extremely ill. Higher scores indicate poor clinical outcome.
Time Frame: At Day 365 (EOT)
Population: CGI-S was assessed and reported for the participant with Dravet Syndrome. As both participants with Tuberous Sclerosis Complex consented under a previous protocol version that did not include CGI S, this assessment was not collected for these participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tuberous Sclerosis Complex | Dravet Syndrome
Number analyzed (Participants) | 0 | 1
score on a scale
  Sensory |  | 3.0 (NA) — Standard deviation cannot be calculated for 1 person.
  Motor |  | 3.0 (NA) — Standard deviation cannot be calculated for 1 person.
  Cognition |  | 4.0 (NA) — Standard deviation cannot be calculated for 1 person.
  Emotional/Behavioral |  | 3.0 (NA) — Standard deviation cannot be calculated for 1 person.
  Communication |  | 4.0 (NA) — Standard deviation cannot be calculated for 1 person.
  Social |  | 1.0 (NA) — Standard deviation cannot be calculated for 1 person.
  Adaptive Functioning |  | 1.0 (NA) — Standard deviation cannot be calculated for 1 person.

19. Primary Outcome: Clinician Global Impression of Change (CGI/C) Score
Description: The CGI/C is a comprehensive neurodevelopmental assessment that covers the following domains: sensory, motor, cognition, emotional/behavioral health, communication, social, and adaptive functioning. This assessment is a 2-question survey per domain to be completed by the clinician. Individual domain scores are reported.
  The severity of impairment in each domain is rated by the clinician in a scale of 1 through 7 where 1 = Normal, not at all ill; 2 = Borderline ill; 3 = Mildly ill; 4 = Moderately ill; 5 = Markedly ill; 6 = Severely ill; 7 = Among the most extremely ill. Higher scores indicate poor clinical outcome.
Time Frame: At Day 365 (EOT)
Population: CGI-C was assessed and reported for the participant with Dravet Syndrome. As both participants with Tuberous Sclerosis Complex consented under a previous protocol version that did not include CGI-C, this assessment was not collected for these participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tuberous Sclerosis Complex | Dravet Syndrome
Number analyzed (Participants) | 0 | 1
score on a scale
  Sensory |  | 3.0 (NA) — Standard deviation cannot be calculated for 1 person.
  Motor |  | 3.0 (NA) — Standard deviation cannot be calculated for 1 person.
  Cognition |  | 3.0 (NA) — Standard deviation cannot be calculated for 1 person.
  Emotional/Behavioral |  | 3.0 (NA) — Standard deviation cannot be calculated for 1 person.
  Communication |  | 4.0 (NA) — Standard deviation cannot be calculated for 1 person.
  Social |  | 3.0 (NA) — Standard deviation cannot be calculated for 1 person.
  Adaptive Functioning |  | 4.0 (NA) — Standard deviation cannot be calculated for 1 person.

20. Other Pre Specified Outcome: Infant and Toddler Quality of Life Questionnaire Short Form 47 (ITQOL-47) Score
Description: The Infant and Toddler Quality of Life Questionnaire Short Form 47 (ITQOL-47) was developed for use in infants and toddlers from 12-months-to-5 years of age and assesses levels of health and well-being. The caregiver will complete the assessment on an electronic device. For each concept, item responses are scored, summed, and transformed on a scale from 0 (worst health) to 100 (best health). Higher scores indicate better clinical outcome.
Time Frame: At Day 365 (EOT)
Population: ITQOL-47 score was assessed in participants with available data in the Safety Analysis Set.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tuberous Sclerosis Complex | Dravet Syndrome
Number analyzed (Participants) | 1 | 1
score on a scale
  Bodily Pain/Discomfort Zone | 0 (NA) — Standard deviation cannot be calculated on 1 person. | 12.50 (NA) — Standard deviation cannot be calculated on 1 person.
  Combined Behavior Scale | 17.90 (NA) — Standard deviation cannot be calculated on 1 person. | 0 (NA) — Standard deviation cannot be calculated on 1 person.
  Change in Health Score | 0 (NA) — Standard deviation cannot be calculated on 1 person. | 1.0 (NA) — Standard deviation cannot be calculated on 1 person.
  Family Cohesion Score | -55.0 (NA) — Standard deviation cannot be calculated on 1 person. | 15.0 (NA) — Standard deviation cannot be calculated on 1 person.
  Growth and Development Score | 5.0 (NA) — Standard deviation cannot be calculated on 1 person. | -15.0 (NA) — Standard deviation cannot be calculated on 1 person.
  General Health Perceptions Score | -20.0 (NA) — Standard deviation cannot be calculated on 1 person. | -20.0 (NA) — Standard deviation cannot be calculated on 1 person.
  Overall Health Score | 25.0 (NA) — Standard deviation cannot be calculated on 1 person. | 0 (NA) — Standard deviation cannot be calculated on 1 person.
  Physical Abilities Score | 11.10 (NA) — Standard deviation cannot be calculated on 1 person. | -5.60 (NA) — Standard deviation cannot be calculated on 1 person.
  Parental Impact-Emotional Score | -25.00 (NA) — Standard deviation cannot be calculated on 1 person. | 12.50 (NA) — Standard deviation cannot be calculated on 1 person.
  Parental Impact-Time Score | 0 (NA) — Standard deviation cannot be calculated on 1 person. | 8.30 (NA) — Standard deviation cannot be calculated on 1 person.
  Temperament and Moods Score | -8.30 (NA) — Standard deviation cannot be calculated on 1 person. | 4.20 (NA) — Standard deviation cannot be calculated on 1 person.

21. Secondary Outcome: Number of Treatment Responders
Description: Treatment Responders are defined as participants with ≥ 50% reduction from baseline in caregiver-reported total countable seizures
Time Frame: Day 1 up to the taper period, up to Week 52
Population: Treatment response was assessed and reported for participants with available data. The participant with Dravet Syndrome was not assessed at the last 3 timepoints due to early withdrawal from the study.
Measure: Number; unit: participants
Arm/Group | Tuberous Sclerosis Complex | Dravet Syndrome
Number analyzed (Participants) | 2 | 1
participants
  Day 1-29 | 0 | 0
  Day 30-57: number analyzed (Participants) | 1 | 1
  Day 30-57 | 0 | 1
  Day 58-85: number analyzed (Participants) | 1 | 1
  Day 58-85 | 0 | 1
  Day 86-113: number analyzed (Participants) | 1 | 1
  Day 86-113 | 1 | 1
  Day 114-141: number analyzed (Participants) | 1 | 1
  Day 114-141 | 1 | 1
  Day 142-169: number analyzed (Participants) | 1 | 0
  Day 142-169 | 1 |
  Day 170-197: number analyzed (Participants) | 1 | 0
  Day 170-197 | 1 |
  Taper Period: number analyzed (Participants) | 1 | 0
  Taper Period | 0 |

22. Other Pre Specified Outcome: Percentage Change From Baseline in Indication-Specific Seizure Frequency As Recorded by Caregivers
Time Frame: Day 1 up to Taper Period, up to Week 52
Population: Seizure frequency was assessed in participants with available data in the Safety Analysis Set.
Measure: Mean (Standard Deviation); unit: seizure frequency
Arm/Group | Tuberous Sclerosis Complex | Dravet Syndrome
Number analyzed (Participants) | 2 | 1
seizure frequency
  Day 1-29 | 56.05 (26.23) | -67.80 (NA) — Standard deviation cannot be calculated for 1 person.
  Day 30-57: number analyzed (Participants) | 1 | 1
  Day 30-57 | 24.80 (NA) — Standard deviation cannot be calculated for 1 person. | -89.50 (NA) — Standard deviation cannot be calculated for 1 person.
  Day 58-85: number analyzed (Participants) | 1 | 1
  Day 58-85 | 2.70 (NA) — Standard deviation cannot be calculated for 1 person. | -94.70 (NA) — Standard deviation cannot be calculated for 1 person.
  Day 86-113: number analyzed (Participants) | 1 | 1
  Day 86-113 | -95.20 (NA) — Standard deviation cannot be calculated for 1 person. | -80.20 (NA) — Standard deviation cannot be calculated for 1 person.
  Day 114-141: number analyzed (Participants) | 1 | 1
  Day 114-141 | -97.60 (NA) — Standard deviation cannot be calculated for 1 person. | -85.80 (NA) — Standard deviation cannot be calculated for 1 person.
  Day 142-169: number analyzed (Participants) | 1 | 0
  Day 142-169 | -97.80 (NA) — Standard deviation cannot be calculated for 1 person. |
  Day 170-197: number analyzed (Participants) | 1 | 0
  Day 170-197 | -88.10 (NA) — Standard deviation cannot be calculated for 1 person. |
  Taper Period: number analyzed (Participants) | 1 | 0
  Taper Period | 71.90 (NA) — Standard deviation cannot be calculated for 1 person. |

23. Secondary Outcome: Number of Participants Who Achieved Seizure-Free Status
Time Frame: Week 12, and every 4 weeks thereafter, up to date of withdrawal or Week 24, whichever occurs first
Population: Seizure free status is reported for the 2 participants that remained on the study for > 12 weeks, and data are reported up to the timepoint prior to their withdrawal from the study. One participant with Tuberous Sclerosis Complex withdrew from the study prior to week 12 so their seizure free status could not be assessed.
Measure: Number; unit: participants
Arm/Group | Tuberous Sclerosis Complex | Dravet Syndrome
Number analyzed (Participants) | 1 | 1
participants
  Week 12 | 0 | 0
  Week 16 | 0 | 0
  Week 20 | 0 | 0
  Week 24: number analyzed (Participants) | 1 | 0
  Week 24 | 0 |

24. Secondary Outcome: Percentage of Participants Still Receiving GWP42003-P
Time Frame: Week 12, and every 4 weeks thereafter, up to date of withdrawal or Week 24, whichever occurs first
Population: Percentage of participants still receiving GWP42003-P is reported to the point at which subjects terminated their treatment and withdrew from the study. One participant with Tuberous Sclerosis Complex withdrew from the study prior to week 12. One participant with Tuberous Sclerosis Complex withdrew following the Day 170-197 timepoint. The participant with Dravet Syndrome withdrew following the Day 142-169 timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Tuberous Sclerosis Complex | Dravet Syndrome
Number analyzed (Participants) | 2 | 1
percentage of participants
  Week 12 | 50 | 100
  Week 16 | 50 | 100
  Week 20 | 50 | 100
  Week 24 | 50 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline up to 62 weeks.
Arm/Group | Tuberous Sclerosis Complex | Dravet Syndrome
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 2/2 | 0/1
Other Adverse Events (participants affected / at risk) | 1/2 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tuberous Sclerosis Complex (N=2) | Dravet Syndrome (N=1)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 (2) | 0 (0)
Change in seizure presentation (Nervous system disorders) | 2 (5) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tuberous Sclerosis Complex (N=2) | Dravet Syndrome (N=1)
Teething (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (3) | 0 (0)
Rhinovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Three participants were enrolled. There was not enough information to answer the research questions. The limited data collected were not enough to provide meaningful conclusions regarding the efficacy, safety, and PK of CBD-OS in this clinical trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-01-24): https://cdn.clinicaltrials.gov/large-docs/04/NCT04485104/Prot_000.pdf
  • Statistical Analysis Plan (2025-03-04): https://cdn.clinicaltrials.gov/large-docs/04/NCT04485104/SAP_001.pdf